CLINICAL TRIAL: NCT06816082
Title: Internet-based Acceptance Based Psychotherapy As an Adjunct to Chronic Pain Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Nina Bendelin, Lic Psychologist, Clinical Researcher, PhD, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-06790-01
Record Dates: First submitted 2025-01-10; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Pain
Keywords: chronic pain; acceptance and commitment therapy; internet delivered treatment
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Internet delivered acceptance and commitment therapy (Experimental): 7 week long treatment with therapist asynchronous support in mainly text format. Treatment includes for example mindfulness, psychoeducation, values, and self-compassion
  Interventions: Behavioral: Internet delivered acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Internet delivered acceptance and commitment therapy — 7 week long treatment with therapist asynchronous support in mainly text format. Treatment includes for example mindfulness, psychoeducation, values, and self-compassion

SUMMARY:
The goal of this clinical trial is to evaluate how an acceptance based internet-delivered psychological treatment (IACT) tailored to patients with chronic pain is perceived, and if it meets the needs and expectations of those enrolled.

The main question it aims to answer is:

What are the expectations of patients with chronic pain prior to IACT treatment, and how do they experience IACT during and after treatment?

Participants will be offered a 7 week long treatment with therapist support. They will be interviewed before treatment starts, once during treatment, and again after treatment is completed.

DETAILED DESCRIPTION:
This research project aims to interview adults with chronic pain to explore their expectations before, during, and after receiving internet-based Acceptance and Commitment Therapy (IACT). IACT aims to increase accessibility to psychological treatment by overcoming geographical, economic, social, or physical barriers. The study will investigate how IACT is received and how patient expectations align with their treatment experiences. This is important because previous studies have shown that chronic pain patients' experiences with IACT vary greatly, and there is limited knowledge about their specific needs and expectations regarding internet-based psychological treatment.

Chronic pain is a widespread and challenging condition affecting approximately 20% of the population. Internet-delivered psychological treatments, such as IACT, have emerged in the past 20 years, showing promising results in managing chronic pain. However, research on patient expectations and experiences with IACT remains limited. This qualitative study will use semi-structured interviews to gather data from 10-15 adults with chronic pain. Three interviews will be conducted per participant: before, during, and after IACT treatment. Thematic analysis will be used to analyze the interview transcripts.

The IACT treatment will consist of 7 modules delivered over 7 weeks. The study's findings will hopefully contribute to a better understanding of how expectations and needs influence the treatment process and outcomes for individuals with chronic pain receiving IACT. This knowledge can inform the development and delivery of more effective and patient-centered IACT programs.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be adults with sufficient understanding of Swedish to speak and read, have internet access, and currently be a patient at the Pain and Rehabilitation Clinic in Linköping.

Exclusion Criteria:

* Severe cognitive problems, or severe mental illness such as a psychotic episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Main outcome - qualitative | Before treatment starts, once in the middle of treatment (3 weeks after start), and after treatment has ended (at 7 weeks post start).
  Semi-structured interviews with patients experiencing chronic pain will be conducted before, during, and after IACT treatment. The interviews will be analyzed thematically to identify recurring themes related to patients' expectations of IACT treatment, their experiences during the treatment, their perceptions of the treatment, and the extent to which the treatment meets their needs. The main areas that will be explored include, but are not limited to, expectations regarding function, pain perception, and quality of life; experiences of the treatment process; perceived benefits and drawbacks of the treatment; and perceptions of whether the treatment addressed their individual needs.

SECONDARY OUTCOMES:
Quantitative - Brief Pain Inventory | Pre and post (7 weeks)
  The pain interference part of the Swedish version of the Brief Pain Inventory - Short Form. A higher scores indicate greater severity and interference. Min: 0. Max: 70.
Quantitative - Chronic Pain Acceptance Questionnaire 8 | pre and post (7 weeks)
  8 items long acceptance questionnaire with two sub scales. For the Engagement subscale, a higher score indicates more engagement in valued activities. For the pain willingness sub scale, a higher score indicates a greater willingness to experience pain. Min: 0. Max: 48.
Quantitative -Pain Self-Efficacy Questionnaire 8 | pre and post (7 weeks)
  8 item long questionnaire measuring self efficacy. Higher scores indicate greater levels of confidence in dealing with pain. Min: 0. Max: 48.
Quantitative - Pain Catastrophizing Scale | pre and post (7 weeks)
  13 item long questionnaire about pain related catastrophizing with three sub scales. Higher scores indicate a greater degree of pain catastrophizing. Min: 0. Max: 52.
Quantitative - Numeric rating scale | Pre and post (7 weeks)
  Average pain during the last 24 hours, from 0 to 10. Higher scores indicate more pain.
Quantitative -Patient Global Impression of Change | Post only (7 weeks)
  Single question with 7 predetermined answers regarding perceived benefit or deterioration. Lower scores indicate deterioration and higher improvement.
Quantitative - Brunnsviken Brief Quality of Life Scale | Pre and post (7 weeks)
  Short quality of life measure. Higher scores indicate greater quality of life. Min: 11. Max: 77.
Quantitative - Patient Health Questionnaire 9 | Pre and post (7 weeks)
  9 item long depression inventory. Higher scores indicate more depressive symptoms. Min: 0. Max: 27.
Quantitative - Generalized Anxiety Disorder 7 | Pre and post (7 weeks)
  7 items long anxiety inventory. A higher score means more anxiety. Min: 0. Max: 21.
Quantitative - Negative effects questionnaire | Post only (7 weeks)
  20 item long questionnaire to measure negative or unwanted effects of treatment.
  Scoring guide by original authors:
  The self-report measure consists of three parts. First, respondents endorse specific items in case they have occurred or not during treatment, yes/no (dummy coded as a variable: 1/0). Second, the respondents rate how negatively the negative effect was on four-point Likert-scale, ranging from "Not at all" to "Extremely", 0-4 ("0" being minimum and "4" being maximum). Third, the respondents attribute the negative effect to "The treatment I received" (1) or "Other circumstances" (0) (dummy coded as a variable: 1/0).

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bendelin, PhD, Principal Investigator — Region Östergötland
Locations (1):
- Pain and Rehabilitation Clinic, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Might interfere with ethical approval.